CLINICAL TRIAL: NCT03814902
Title: A Prospective Pilot Study to Characterize the Impact on Families of Electronic Tracking Device Use by Children With Autism Spectrum Disorders Who Wander
Brief Title: A Pilot Study to Characterize the Household Impact of Locating Devices for Children With ASD Who Wander
Acronym: CHILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-0314_A
Record Dates: First submitted 2019-01-10; First posted 2019-01-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder; Wandering Behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Wandering Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic Tracking Device (Experimental): Participants will be given a wearable electronic tracking device (ETD) to use for their child with autism spectrum disorder (ASD) for 6 weeks.
  Interventions: Device: Electronic Tracking Device

INTERVENTIONS:
Device: Electronic Tracking Device — This commercially-available electronic tracking device uses Global Positioning System (GPS) technology to display the wearer's location on a mobile phone, tablet, or computer. The device may be securely attached to clothing and is designed to be worn by children with developmental disabilities. Parents may use the associated application to view the child's location when the device is turned on and active.

SUMMARY:
This pilot study will obtain preliminary data about the impact of wearable electronic tracking devices (ETDs) as an intervention for children with autism spectrum disorders (ASD) who wander. The feasibility of all study procedures and the acceptability of the intervention will be evaluated.

DETAILED DESCRIPTION:
Wandering, or elopement, is a life-threatening behavior that has been reported to occur in a third of all children with autism spectrum disorders (ASD). Wearable electronic tracking devices (ETDs) that are able to pinpoint a child's location have emerged as an appealing intervention for families concerned about wandering risk. However, the impact of ETD use on the families of children who wander has never been studied prospectively. In this pilot study, parents will be provided with a commercially-available ETD to use for their child with ASD for 6 weeks. Preliminary data will be obtained to evaluate the impact of ETD use on the strain experienced by families due to their child's wandering behavior. The feasibility of all study procedures will be assessed in preparation for a larger subsequent trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Parent of a child between the ages of 4 and 17 who currently has autism spectrum disorder (ASD), was diagnosed with ASD by a professional, and has wandered at least once in the preceding 3 months
* Currently lives in the United States
* Currently lives with child with ASD
* Has been living with child with ASD for at least 6 months
* Has reliable internet access to allow for completion of online questionnaires

Exclusion Criteria:

Current or past use of any electronic tracking device to address wandering behavior in the child with ASD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Rates of participant retention | 6 weeks
  Participant retention will be assessed to evaluate the feasibility of all study procedures.
Rates of questionnaire completion | 6 weeks
  Questionnaire completion rates will be calculated to assess the feasibility of the proposed evaluation schedule.
Adherence to the intervention | 6 weeks
  The mean daily duration of participant use of the device will be assessed to evaluate the acceptability of the intervention.

SECONDARY OUTCOMES:
Changes from baseline in Caregiver Strain Questionnaire (CGSQ) scores | Baseline and Week 6
  The Caregiver Strain Questionnaire is a validated, 21-item instrument that was developed to measure the strain experienced by parents of children with emotional and behavioral disorders. A modified version of this questionnaire will be administered in order to evaluate parental strain due to wandering-related concerns. The questionnaire measures three dimensions of caregiver strain, including objective strain (11 items), internalized subjective strain (6 items), and externalized subjective strain (4 items). Each subscale score is calculated by averaging responses (on a five-point scale) to all items in the subscale. A global score is obtained by summing all three subscale scores, with higher scores indicating a greater degree of caregiver strain.
Changes from baseline in GAD-7 scores | Baseline, Week 6
  The Generalized Anxiety Disorder 7-Item (GAD-7) scale is a validated measure of the severity of anxiety symptoms. Possible scores range from 0 to 21, with higher scores indicating more severe levels of anxiety.
Changes from baseline in BFDS scores | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  The Brief Family Distress Scale (BFDS) is a single-item measure for evaluating the experience of distress or crisis in families of children with developmental disabilities. Possible scores range from 1 to 10, with higher scores representing a greater degree of family distress.
Changes from baseline in the frequency of wandering-related disruptions to the household. | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  A weekly study-specific questionnaire will evaluate the perceived impact of the child's wandering behavior on parent, child, and family activities.
Perceived impact of the intervention | 6 weeks
  Study-specific questionnaires will assess the perceived impact of the intervention on the child's wandering behavior and on the well-being of the parent and child.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Adesman, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiely B, Migdal TR, Vettam S, Adesman A. Prevalence and Correlates of Elopement in a Nationally Representative Sample of Children with Developmental Disabilities in the United States. PLoS One. 2016 Feb 4;11(2):e0148337. doi: 10.1371/journal.pone.0148337. eCollection 2016. PMID 26845701